CLINICAL TRIAL: NCT04808349
Title: Safety and Efficacy in a ReAl-Life Study in Patients With Haemophilia Treated wIth NovoEight® for Surgery
Acronym: SERAPHINE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0053
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
the aim of the SERAPHINE study is to gather data stemming from the French research database BERHLINGO (= Base d'Etude et de Recherche en Hémostase pour Les Investigateurs du Grand-Ouest, i.e. Database for Research on Hemostasis for the Investigators of Western France), in order to get a detailed report about the therapeutic management and use of turoctocog alfa (NovoEight®) in surgery in pwHA (Patient with inherited Hemophilia A).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Regardless of age
* No inhibitor (anti-FVIII alloantibodies) at the time of treatment.
* No objections expressed to participate in the study after having been informed of its purposes and the data involved.
* No other inherited hemorrhagic disorders than HA

Exclusion Criteria:

In order to reflect the reality of daily practice, no criteria for non-inclusion are provided for other than the refusal of the patient or his or her legal representative to participate in the study or the existence in the patient of a contraindication to the use of turoctocog alfa (NovoEight®) treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to respect the independence of the physicians, this study is conducted with patients for whom the decision to prescribe turoctocog alfa (NovoEight®) treatment is not related to the study. The prescription of turoctocog alfa (NovoEight®) will therefore have been carried out on the initiative of the physicians of the participating centers, in collaboration with the patients involved. This study therefore does not lead to any change in the usual medical care of the people entering the study, nor does it affect the physical or psychological integrity of the patients.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Assessing the effectiveness of turoctocog alfa (NovoEight®) to prevent hemorrhagic complications during minor and major surgery procedures in pwHA | 1 year
  Overall evaluation by the investigator of the hemostatic effectiveness of turoctocog alfa (NovoEight®) for the prevention of hemorrhagic complications in a surgical setting (excellent, good, fair, poor/none according to recommendations of the SSC of ISTH)

SECONDARY OUTCOMES:
Assessing the safety of turoctocog alfa (NovoEight®) when used during surgery in patients with the occurrence of adverse events (AEs), especially hemorrhagic and thrombotic complications or development of inhibitors. | 1 year
  Nature and incidence of AEs, including serious AEs, AEs related to turoctocog alfa (NovoEight®)
Assessing the duration of replacement therapy and factor VIII consumption in clinical practice during surgery in patients treated with turoctocog alfa (NovoEight®) | 1 year
  Number of administrations and total required dose of turoctocog alfa (NovoEight®) in IU/kg

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Angers, Angers
  - CH Le Mans, Le Mans
  - CHU de Nantes, Nantes

IPD SHARING:
Plan to Share IPD: Undecided